CLINICAL TRIAL: NCT06079047
Title: Perineural Dexamethasone in the Adductor Canal Block for Postoperative Pain in Knee Arthroplasty Surgery
Brief Title: Perineural Dexamethasone in the Adductor Canal Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Olfa kaabachi, MD (Other)
Responsible Party: Sponsor-Investigator, Olfa kaabachi, MD, PROFESSOR, University Tunis El Manar
Organization: University Tunis El Manar (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CE-IMKO- 111/2023
Record Dates: First submitted 2023-05-09; First posted 2023-10-12 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2024-02

CONDITIONS: Post Operative Pain
Keywords: knee arthroplasty; glucocorticoids; adductor canal block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group Dexamethasone (Experimental): adductor canal block with 10 ml of 0.5% "bupivacaine" + 10 ml of 0.9% saline solution + 2 ml of "dexamethasone" (8 mg)
  Interventions: Procedure: group Dexamethasone
- group Controle (Active Comparator): adductor canal block with 10 ml of 0.5% "bupivacaine" + 10 ml of 0.9% saline solution + 2 ml of 0.9% saline solution
  Interventions: Procedure: group Controle

INTERVENTIONS:
Procedure: group Dexamethasone — Adductor canal block with dexamethasone
  Arms: group Dexamethasone
Procedure: group Controle — Adductor canal block with saline solution
  Arms: group Controle

SUMMARY:
Postoperative pain management in total knee arthroplasty (TKA) surgery is a real challenge for the anesthesiologist. Effective pain control must be provided while preserving the mobility to ensure early rehabilitation. The adductor canal block is an effective way to induce sensory block without motor block. However, the major disadvantage of this block is the duration of sensory block which may be insufficient for postoperative pain management in TKA surgery. Many studies have focused on finding molecules that can prolong sensory block without the need for a perineural catheter and dexamethasone is among the most studied molecules(1, 2). Hence, our study aims to evaluate the added value of perineural dexamethasone in the adductor canal block in TKA surgery.

[

DETAILED DESCRIPTION:
Using a computer-generated sequence of random numbers, the patients included will be randomly allocated to get an adductor canal block using :

Group D: 10 ml of 0.5% bupivacaine + 10 ml of 0.9% normal saline solution + 8 mg of dexamethasone (equivalent to 2 ml) Group C: 10 ml of 0.5% bupivacaine + 10 ml of 0.9% normal saline solution + 2 ml of 0.9% normal saline solution

All patients included in the study will initially be evaluated at the anesthesia outpatient clinic with correction of any existing health issues. A pre-anesthesia visit will be conducted the day before the procedure for all patients, providing them with information about the protocol of our study and obtaining their consent to participate.

Upon arrival at the operating room, non-invasive monitoring of blood pressure, pulse oximetry, and ECG tracing will be performed and also a blood glucose level measurement. An 18-gauge peripheral intravenous line will be established, and 0.03 mg per kg midazolam was administrated.

All patients will receive spinal anesthesia. Depending on the patient's condition, investigators will opte for:

A single shot spinal anesthesia using 0.5% bupivacaine (11 mg) with fentanyl (25 µg) for patients under 65 years of age with ASA I and II Continuous spinal anesthesia with drug titration for patients over 65 years of age or with ASA III classification.

None of patients will receive intravenous dexamethasone during the perioperative period.

The decision to use a tourniquet and use of cement will be left to the surgeon. In the immediate postoperative period, all patients will receive an adductor canal block with a high-frequency probe. The patients will be positioned in a supine position with the leg slightly externally rotated. The probe will be placed transversely on the inguinal fold. The femoral vessels (artery and vein) will be identified. The different muscular structures delimiting the adductor canal will be visualized: the sartorius muscle that covers the femoral artery and the medial vastus muscle laterally. The saphenous nerve, which is usually hyperechoic, is located most often at the lateral edge of the artery in the fascia between the sartorius and medial vastus muscles. A 100 mm neurostimulation needle was used and 22 ml solution was injected into the adductor canal.

Patients will be transferred to continuous care unit for 48 hours.

Post operative analgesia will include:

1. Paracetamol 1g IV every 6 hours for 1 day then oral paracetamol 1g every 8 hours for 4 weeks
2. Diclofenac sodium (50 mg) *2 per day for 5 days
3. PCA morphine (Patient Controlled Analgesia), as a rescue analgesia. The first rise will be allowed on day 1 (18 h postoperatively) and the patient will be asked to wander with a walking frame for a distance of at least 3 meters (about 10 steps).

The patient will be considered ready for discharge after completing protocol endpoints and walking at least 3 meters without support.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for unilateral TKA
* Surgery under spinal anesthesia
* ASA class I, II, and III patients

Exclusion Criteria:

* Patient refusal to participate in the study
* Contraindication to regional anesthesia
* Allergies to the products used
* Bilateral TKA
* Revision TKA
* TKA in the context of inflammatory or post-traumatic disease
* BMI > 45
* Poorly controlled diabetic patients with HbA1c > 8%
* Patients on corticosteroid therapy or who have received an intra-articular injection of corticosteroids

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2023-12-15 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
morphine consumption | 48 hours
  postoperative consumption of morphine

SECONDARY OUTCOMES:
NRS at rest | 1 hour, 3 hours, 6 hours, 9 hours,12 hours, 24 hours, 36 hours and 48 hours postoperatively
  Numerical rate scale at rest [ NRS =0 no pain ; NRS =10 worse pain]
NRS on mouvement | 1 hour, 3 hous, 6 hours, 9 hours,12 hours, 24 hours, 36 houes and 48 hours postoperatively
  Numerical rate scale during knee flexion [ NRS =0 no pain ; NRS =10 worse pain]
knee mouvement | preoperatively, on day 1 and day 7 postoperatively
  Range of mouvement of the knee
walk | day 1 and day 2 postoperatively
  Numbers of steps
Patient's satisfaction | 48 hours postoperatively
  3 level scale :0: not satisfied; 1: mild satisfaction; 2: satisfied
Blood glucose level | 1 hour, 6 hours,12 hours,18 hours, 24 hours postoperatively
  Blood glucose level
pain at home | 7 days postoperatively
  NRS at mouvement [ NRS =0 no pain ; NRS =10 worsE pain]
quality of recovery | day one
  QoR15 score [ 136-150 excellent recovery - 0-89 poor recovery]
neuropathic Chronic pain | 6 MONTHS
  DN4 questionnaire [ no neuropathic pain 0 - neuropathic pain >4]
chronic pain | 6 months
  NRS on mouvement [ NRS =0 no pain ; NRS =10 worse pain]
postoperative quality of life | 6 months
  SF-12 score [0 to 100, with higher scores indicating better physical and mental health functioning]
knee fonction | 6 months
  KOOS PS score [[0 to 100, with higher scores indicating better knee function]functioning]

CONTACTS AND LOCATIONS:
Locations (1):
- KAABACHI, Tunis, La Mannouba, Tunisia

IPD SHARING:
Plan to Share IPD: No